CLINICAL TRIAL: NCT00390689
Title: A Randomised, Double-blind Study to Evaluate the Efficacy and Safety of Pramipexole at Fixed Doses of 0.25 mg, 0.5 mg, and 0.75 mg in Patients With Idiopathic Restless Legs Syndrome for 6 Weeks, Followed by a 46-week Open-label Long-term Study
Brief Title: A Randomised, Comparing Fixed Doses of Pramipexole to Investigate the Efficacy and Safety in Patients With RLS.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.627
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-04

CONDITIONS: Idiopathic Restless Legs Syndrome
MeSH Terms: interventions — Pramipexole; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Pramipexole 0.25 mg once daily (Experimental): Pramipexole 0.25 mg given once daily
  Interventions: Drug: Pramipexole 0.125 mg tablet
- Pramipexole 0.5 mg once daily (Experimental): Pramipexole 0.5 mg given once daily
  Interventions: Drug: Pramipexole 0.5 mg tablet
- Pramipexole 0.75 mg once daily (Experimental): Pramipexole 0.75 mg given once daily
  Interventions: Drug: Pramipexole 0.125 mg tablet; Drug: Pramipexole 0.5 mg tablet

INTERVENTIONS:
Drug: Pramipexole 0.125 mg tablet
  Arms: Pramipexole 0.25 mg once daily; Pramipexole 0.75 mg once daily
Drug: Pramipexole 0.5 mg tablet
  Arms: Pramipexole 0.5 mg once daily; Pramipexole 0.75 mg once daily

SUMMARY:
The objective of double blind phase in this trial is to compare the efficacy and safety at the fixed dose of 0.25 mg,0.5 mg and 0.75 mg pramipexole in RLS. The objective of open label phase in this trial is to investigate the long term safety and efficacy of pramipexole in RLS.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 20 and 80 years
2. Patients with a diagnosis of restless legs syndrome (RLS) according to the following diagnosis criteria of National institute of health (NIH)/International restless legs syndrome study group (IRLSSG):

   1. An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs.
   2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying or sitting.
   3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
   4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night.
3. Patients with a total score larger than 15 on the IRLS at Visit 2

Exclusion Criteria:

1. Premenopausal women who meet any of the following 1) to 3) 1) Patients who are pregnant or possibly pregnant 2) Patients who are lactating 3) Patients who wish to become pregnant during the study period
2. Patients who cannot take adequate contraceptive measures
3. Patients with a history of akathisia induced by neuroleptics
4. Patients with diabetes mellitus requiring insulin therapy
5. Patients who are judged to have microcytic anaemia by the investigator or sub-investigator
6. Patients with a history or signs of peripheral neuropathy, myelopathy, multiple sclerosis, Parkinson's disease or other neurological diseases that may result in the occurrence of secondary RLS in the physical function tests or neurological tests
7. Patients with other sleep disorders such as abnormal behaviour during Rapid eye movement (REM) sleep, narcolepsy and sleep apnoea syndrome (patients with an apnoea-hypopnoea index (AHI) exceeding 15 determined by polysomnography at the relevant trial site or those with loud snoring at least 5 nights/week and an experience of respiratory arrest during sleep or excessive daytime sleepiness)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (34):
- Japan (34):
  - 248.627.037 Boehringer Ingelheim Investigational Site, Aichi-gun, Aichi
  - 248.627.014 Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - 248.627.029 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 248.627.032 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 248.627.030 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 248.627.013 Boehringer Ingelheim Investigational Site, Kanagawa, Yokohama
  - 248.627.033 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 248.627.027 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 248.627.023 Boehringer Ingelheim Investigational Site, Kitakyusyu, Fukuoka
  - 248.627.024 Boehringer Ingelheim Investigational Site, Kitakyusyu, Fukuoka
  - 248.627.022 Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - 248.627.034 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 248.627.038 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 248.627.041 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 248.627.039 Boehringer Ingelheim Investigational Site, Kumamoto, Kumamoto
  - 248.627.003 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 248.627.036 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 248.627.025 Boehringer Ingelheim Investigational Site, Mitaka-shi, Tokyo
  - 248.627.015 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 248.627.017 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 248.627.011 Boehringer Ingelheim Investigational Site, Otaru, Hokkaido
  - 248.627.026 Boehringer Ingelheim Investigational Site, Otsu, Shiga
  - 248.627.002 Boehringer Ingelheim Investigational Site, Sakai,Osaka
  - 248.627.010 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 248.627.035 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 248.627.012 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 248.627.001 Boehringer Ingelheim Investigational Site, Shibuya-ku, Tokyo
  - 248.627.004 Boehringer Ingelheim Investigational Site, Shimotsuga-gun,Tochigi
  - 248.627.040 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 248.627.018 Boehringer Ingelheim Investigational Site, Takatsuki,Osaka
  - 248.627.028 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 248.627.019 Boehringer Ingelheim Investigational Site, Tokushima, Tokushima
  - 248.627.016 Boehringer Ingelheim Investigational Site, Toyohashi, Aichi
  - 248.627.031 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole 0.25mg Group: Double-blind period: 0.25 mg randomised group
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 2 tablets of 0.125mg Pramipexole + 2 tablets of the matching placebo once daily Week 4-6: 2 tablets of 0.125mg Pramipexole + 4 tablets of the matching placebo once daily
  Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.5mg Group: Double-blind period: 0.5 mg randomised group
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 4 tablets of 0.125mg Pramipexole once daily Week 4-6: 4 tablets of 0.125mg Pramipexole + 2 tablets of the matching placebo once daily
  Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.75mg Group: Double-blind period: 0.75 mg randomised group
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 4 tablets of 0.125mg Pramipexole once daily Week 4-6: 6 tablets of 0.125mg Pramipexole once daily
  Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  mode of administration.: Oral, once daily, 2-3 hours before bedtime
Period: Overall Study
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Started | 48 | 53 | 53
Completed | 43 | 48 | 50
Not Completed | 5 | 5 | 3
Not completed — Adverse Event | 2 | 5 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Investigator's judgement | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group | Total
Number analyzed (Participants) | 48 | 53 | 53 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.9) | 52.4 (12.9) | 54.3 (14.4) | 53.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 32 | 89
  Male | 18 | 26 | 21 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Restless Legs Syndrome (IRLS) Total Score at 6 Weeks
Description: The International Restless Legs Syndrome Study Group (IRLSSG) proposes classification of severity based on the total score on the IRLS (0-10, mild; 11-20, moderate; 21-30, severe; 31-40, very severe). A decrease in the score of the IRLS by 10 or more points corresponds to the improvement of severity by one rank and has clinical importance. Therefore, the primary endpoint in the double-blind period was set as a decrease by 10 or more points in the mean change on the total score of the IRLS from the baseline to Visit 5 (last observation day in the double-blind period) at all doses of 0.25 mg, 0.5 mg, and 0.75 mg/day of pramipexole.
Time Frame: Week 6 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
Points on a scale | -12.3 (1.1) | -12.5 (1.1) | -11.8 (1.1)

2. Secondary Outcome: IRLS Responder
Description: The percentage of patients with 50 % or more reduction of IRLS (The measure means the percentage of high responder on the trial medications)
Time Frame: baseline to week 6
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
Percentage of patients | 60.4 | 58.5 | 49.1

3. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Score at 6 Weeks
Description: PSQI developed to evaluate the quality of sleep is a self-recording questionnaire consisting of 18 questions focused on 7 factors such as sleep quality, sleep period time, sleep latency, sleep efficiency, sleep difficulty, use of hypnotics, and hindrance to activities of daily living due to daytime sleepiness. Each score (0-3 points) in the respective factors was added to calculate the total score (0-21 points). Rating scale scored from 0 (best sleep) to 21 (worst sleep).
Time Frame: Week 6 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 46 | 50 | 48
Points on a scale | -3.2 (0.4) | -3.2 (0.4) | -2.5 (0.4)

4. Secondary Outcome: Change From Baseline in Japanese Version of the Epworth Sleepiness Scale (JESS) Total Score at 6 Weeks
Description: ESS is a self-recording scale used to evaluate sleepiness experienced in daily activities and it consists of 8 items focused on specific situations such as reading books and watching television. Each score (0-3 points) to 8 questions was added simply to calculate the total ESS score. A Japanese translation of the ESS (a provisional version provided by the Japanese Respiratory Society) used so far had not been prepared through the international scale development and validation process, but the version prepared through this process was published at the 31st meeting of the Japanese Society of Sleep Research. The questions in JESS had been discussed with the original author of the ESS and their measurement concepts had been confirmed. The JESS is the Japanese version of ESS prepared through the international scale development and validation process. Rating scale scored from 0 (no daytime sleep) to 24 (worst daytime sleep)
Time Frame: Week 6 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
Points on a scale | -2.6 (0.6) | -3.0 (0.5) | -2.3 (0.6)

5. Secondary Outcome: Clinical Global Impression Global Improvement (CGI-I) Responder
Description: CGI is extensively used for risk-benefit evaluation (efficacy) of drug therapies. The CGI evaluates the severity and improvement in 7 ranks. It also evaluates the therapeutic effect and side effects in 4 ranks, separately. Rating scale from 1 (very much improved) to 7 (very much worse). The percentage of patients who were evaluated as 1(very much improved) or 2(much improved) by the investigator were considered responders.
Time Frame: baseline to week 6
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
Percentage of patients | 77.1 | 75.5 | 69.8

6. Secondary Outcome: Patient Global Impression (PGI) Responder
Description: PGI is used to evaluate a global impression by patients themselves in 7 ranks. Rating scale from 1 (very much better) to 7 (very much worse). The percentage of patients where the patient evaluated himself/herself as 1(very much better) or 2(much better)were considered responders.
Time Frame: baseline to week 6
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
Percentage of patients | 72.9 | 79.2 | 67.9

7. Secondary Outcome: Clinically Significant Abnormalities in Vital Signs (Blood Pressure and Pulse Rate in Both Supine and Standing Positions), ECG, Laboratory Tests - Double Blind Period.
Time Frame: baseline to 6 weeks
Measure: Number; unit: participants
Arm/Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 48 | 53 | 53
participants
  Blood pressure increased | 0 | 1 | 0
  Cardiovascular disorder | 0 | 0 | 1

8. Secondary Outcome: Change From Baseline in International Restless Legs Syndrome (IRLS) Total Score at 52 Weeks for Open-Label Period
Description: The International Restless Legs Syndrome Study Group (IRLSSG) proposes classification of severity based on the total score on the IRLS (0-10, mild; 11-20, moderate; 21-30, severe; 31-40, very severe).
Time Frame: Week 52 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Pramipexole 0.125mg Group: Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.125 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.25mg Group: Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.25 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.5mg Group: Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.5 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.75mg Group: Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.75 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Points on a scale | -18.5 (5.8) | -17.3 (5.8) | -18.3 (6.1) | -14.8 (8.9)

9. Secondary Outcome: IRLS Responder for Open-label Period
Description: as for outcome 2
Time Frame: baseline to week 52
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Groups:
- Pramipexole 0.50mg Group: Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.5 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.50mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Percentage of patients | 100.0 | 90.0 | 92.0 | 68.0

10. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Total Score at 52 Weeks for Open-Label Period
Description: as for outcome 3
Time Frame: Week 52 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 39 | 49 | 25
Points on a scale | -4.0 (2.4) | -3.3 (3.3) | -3.3 (3.3) | -2.4 (3.8)

11. Secondary Outcome: Change From Baseline in Japanese Version of the Epworth Sleepiness Scale (JESS) Total Score at 52 Weeks for Open-Label Period
Description: as for outcome 4
Time Frame: Week 52 - change from baseline
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Points on a scale | -9.5 (2.9) | -3.8 (4.3) | -4.4 (4.7) | -2.6 (5.7)

12. Secondary Outcome: Clinical Global Impression Global Improvement (CGI-I) Responder at 52 Weeks for Open-label Period
Description: as for outcome 5
Time Frame: baseline to week 52
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Percentage of patients | 100.0 | 95.0 | 98.0 | 84.0

13. Secondary Outcome: Patient Global Impression (PGI) Responder at 52 Weeks for Open-Label Period
Description: as for outcome 6
Time Frame: baseline to week 52
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Percentage of patients | 100.0 | 97.5 | 94.0 | 80.0

14. Secondary Outcome: Possible Augmentation in RLS Symptoms at 52 Weeks for Open-Label Period
Description: Possible augmentation defined as persistence of a state in which RLS symptoms begin to occur 2 hours earlier than the usual time zone for 5 days or more a week
Time Frame: baseline to week 52
Population: Full Analysis Set (FAS).
Measure: Number; unit: Percentage of patients
Arm/Group | Pramipexole 0.125mg Group | Pramipexole 0.25mg Group | Pramipexole 0.5mg Group | Pramipexole 0.75mg Group
Number analyzed (Participants) | 4 | 40 | 50 | 25
Percentage of patients | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication onwards through the observational phase (52 weeks).
Groups:
- Pramipexole 0.25mg (Double-blind): Double-blind period: 0.25 mg randomised group.
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 2 tablets of 0.125mg Pramipexole + 2 tablets of the matching placebo once daily Week 4-6: 2 tablets of 0.125mg Pramipexole + 4 tablets of the matching placebo once daily
- Pramipexole 0.50mg (Double-blind): Double-blind period: 0.5 mg randomised group
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 4 tablets of 0.125mg Pramipexole once daily Week 4-6: 4 tablets of 0.125mg Pramipexole + 2 tablets of the matching placebo once daily
- Pramipexole 0.75mg (Double-blind): Double-blind period: 0.75 mg randomised group
  Administration as follows:
  Week 1: 1 tablet of 0.125mg Pramipexole once daily Week 2: 2 tablets of 0.125mg Pramipexole once daily Week 3: 4 tablets of 0.125mg Pramipexole once daily Week 4-6: 6 tablets of 0.125mg Pramipexole once daily
- Pramipexole 0.125mg (Open Label): Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.125 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.25mg (Open Label): Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.25 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.50mg (Open Label): Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.5 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
- Pramipexole 0.75mg (Open Label): Open-label period:
  Administration of pramipexole was started at 0.25 mg/day at Week 6 (Visit 5, the last observation day in the double-blind period). Subsequently, the Patient Global Impression (PGI) and tolerability was assessed from Visit 6 and if required, the investigator or subinvestigator determined whether to increase the daily dose to 0.5 mg and then to 0.75 mg/day every two weeks. After checking the PGI and tolerability at each visit, the investigator or sub-investigator determined dose increase, maintenance or reduction.
  The end-of-trial dosage was 0.75 mg. mode of administration.: Oral, once daily, 2-3 hours before bedtime
Arm/Group | Pramipexole 0.25mg (Double-blind) | Pramipexole 0.50mg (Double-blind) | Pramipexole 0.75mg (Double-blind) | Pramipexole 0.125mg (Open Label) | Pramipexole 0.25mg (Open Label) | Pramipexole 0.50mg (Open Label) | Pramipexole 0.75mg (Open Label)
Serious Adverse Events (participants affected / at risk) | 0/48 | 2/53 | 0/53 | 1/8 | 5/140 | 0/97 | 0/41
Other Adverse Events (participants affected / at risk) | 32/48 | 42/53 | 42/53 | 5/8 | 58/140 | 50/97 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole 0.25mg (Double-blind) (N=48) | Pramipexole 0.50mg (Double-blind) (N=53) | Pramipexole 0.75mg (Double-blind) (N=53) | Pramipexole 0.125mg (Open Label) (N=8) | Pramipexole 0.25mg (Open Label) (N=140) | Pramipexole 0.50mg (Open Label) (N=97) | Pramipexole 0.75mg (Open Label) (N=41)
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole 0.25mg (Double-blind) (N=48) | Pramipexole 0.50mg (Double-blind) (N=53) | Pramipexole 0.75mg (Double-blind) (N=53) | Pramipexole 0.125mg (Open Label) (N=8) | Pramipexole 0.25mg (Open Label) (N=140) | Pramipexole 0.50mg (Open Label) (N=97) | Pramipexole 0.75mg (Open Label) (N=41)
Nasopharyngitis (Infections and infestations) | 6 | 13 | 6 | 4 | 32 | 29 | 14
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 4 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 4 | 1 | 2 | 5 | 1
Headache (Nervous system disorders) | 5 | 10 | 2 | 0 | 11 | 4 | 3
Somnolence (Nervous system disorders) | 10 | 15 | 9 | 0 | 9 | 11 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eustachian tube stenosis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 3 | 1 | 0 | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 3 | 3 | 0 | 4 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 22 | 25 | 1 | 11 | 15 | 11
Stomach discomfort (Gastrointestinal disorders) | 2 | 4 | 4 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 5 | 1 | 3 | 5 | 4
Abdomial pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 2 | 2
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 2
Thirst (General disorders) | 0 | 2 | 4 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.